CLINICAL TRIAL: NCT04265131
Title: Emotion Regulation in Eating Disorders: How Can Art Therapy Contribute to Treatment Outcome? A Feasibility Study
Brief Title: Emotion Regulation in Eating Disorders: How Can Art Therapy Contribute to Treatment Outcome?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/2019/0785
Record Dates: First submitted 2019-12-05; First posted 2020-02-11 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder
Keywords: art therapy; emotion regulation; treatment
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Emotional Regulation | interventions — Art Therapy

STUDY DESIGN:
Intervention Model Description: The participants are consecutively assigned in two conditions: a within-subjects design. Those from the experimental group receive standard treatment (TAU) with AT as an extra variable. AT is an experiential form of therapy in which art techniques and supplies (including drawing, painting, clay, etc.) are used methodically with a therapeutic purpose. TAU means that individual verbal therapy takes place on a regular basis, whereby the frequency varies depending on the severity of the eating disorder and the patient's request for help. Cognitive-behavioral therapy is provided with elements of dialectical behavioral therapy, and there is also the possibility of family or couple counseling by a family-based therapist. The participants in the control group only receive this standard treatment (TAU), without AT. Waves will be used: a control group will also become an experimental group at a later stage.
  In this way the investigators can investigate the additional added value of AT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): art therapy is delivered on top of treatment as usual (TAU). TAU means that individual verbal therapy takes place on a regular basis, whereby the frequency varies depending on the severity of the eating disorder and the patient's request for help. Cognitive-behavioral therapy is provided with elements of dialectical behavioral therapy, and there is also the possibility of family or couple counseling by a family-based therapist.
  Interventions: Other: art therapy

INTERVENTIONS:
Other: art therapy — Art therapy is a form of psychotherapy that uses creative methods of expression through art media, such as pencils, clay, paint etc.

SUMMARY:
Eating disorders are difficult to treat. Some forms of treatment have already been found to be effective, nevertheless chronicity is a major problem. For example, both cognitive behavioral therapy and family therapy (FBT; family-based treatment) appear to be effective treatment methods, in which FBT distinguishes itself primarily in its long-term effect. However, eating disorders persist in 20 to 25 percent of cases, only 46 percent of patients with Anorexia Nervosa fully recover and one third only partially improve. Since the mortality rate of this mental disorder is particularly high, it is necessary to keep looking to improve treatment. Because emotion regulation problems play an important role in the cause and maintenance of an eating disorder, more emotion-focused therapies may improve treatment outcome. Dialectical Behavioral Therapy is a treatment that has a strong focus on emotions regulation, but so far only limited evidence has been found for the effectiveness of this type of therapy in eating disorders. Some studies show that art therapy (AT; art therapy) can contribute to a more adaptive regulation of emotions. However, this type of therapy has not been studied in the context of eating disorders yet. AT is an experiential form of therapy in which art techniques and supplies (including drawing, painting, clay, etc.) are used methodically with a therapeutic purpose. The idea that creative expression can perpetuate or improve mental well-being has been accepted worldwide for many years. Despite the long history of practical applications, to date little evidence exist on the effectiveness of this form of treatment. There's growing worldwide interest in scientific research and the emphasis on evidence-based practice (EBP) for this form of treatment. In a recent study, Lock and colleagues compare AT with cognitive remediation therapy (CRT) and the added value of both in a sample of adolescents with anorexia nervosa combines with obsessive-compulsive problems. Both CRT and AT are offered in this study in combination with family based therapy (FBT). The group in which the combination of FBT and AT was offered yielded better results than those in which FBT is combined with CRT.

Study hypothesis: the investigators expect that complementing treatment as usual (TAU) with art therapy (AT) will lead to a decrease in emotion regulation problems in patients with an eating disorder in comparison with TAU only, without AT.

ELIGIBILITY:
Inclusion Criteria:

* The participant is diagnosed with an eating disorder by a psychiatrist at the outpatient department of Ghent University Hospital Eating Disorders.
* At the start of the study, the participant is being treated by a psychiatrist or psychologist at the outpatient department of Eating Disorders at UZ Gent.
* The participant is informed about the purpose of the research and informed consent.

Exclusion Criteria:

* The candidate has already had a hospitalization and so art therapy at the eating disorders department at UZ Gent.
* Lower intelligence with an estimated IQ score lower than 85- The candidate participant is a minor at the start of the study.
* The candidate is struggling with a psychotic problem, as determined by the treating physician or psychologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Difficulties in Emotion Regulation Outcome Measures | The outcome measure will be assessed in phase 1= baseline outcome, phase 2= 6 weeks after baseline , phase 3 = 3 weeks after phase 2, phase 4= 3 weeks after phase 3 and phase 5 = 6 weeks after phase 4
  Measured with "Difficulties in Emotion Regulation Scale" (DERS). This questionnaire contains 36 items that are surveyed on 6 different subscales for clinically relevant emotion regulation problems. Items are scored on a five-point scale from 1 (almost never) to 5 (almost always).
Change in Cognitive Emotion Regulation | phase 1= baseline outcome, phase 2= 6 weeks after phase 1, phase 3 = 3 weeks after phase 2, phase 4= 3 weeks after phase 3 and phase 5 = 6 weeks after phase 4
  Measured with Cognitive Emotion Regulation Questionnaire (CERQ). This questionnaire with 36 items, in which is assessed what someone thinks in stressful situations.
Change in the the psychological background of the eating disorder. | phase 1= baseline outcome, phase 2= 6 weeks after phase 1, phase 4= 6 weeks after phase 2 and phase 5 = 6 weeks after phase 4
  Measures with Eating disorder inventory-3 (EDI-3). This self-report questionnaire consists of 2 parts. On the one hand a diagnosis list, based on the DSM-5, on the other hand questions regarding the psychological background of eating disorder.
Change in emotion regulation in art therapy. | phase 3 (=9 weeks after baseline outcome measure outcome 1,2 and 3) and phase 4= 3 weeks after phase 3
  Measures with "Expression And Emotion Regulation in Art Therapy Scale" (SERATS) This is a short questionnaire with 9 items asking for emotion regulation in art therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Belgium

REFERENCES:
- [Background] Fairburn CG, Harrison PJ. Eating disorders. Lancet. 2003 Feb 1;361(9355):407-16. doi: 10.1016/S0140-6736(03)12378-1. PMID 12573387
- [Background] Juarascio A, Shaw J, Forman E, Timko CA, Herbert J, Butryn M, Bunnell D, Matteucci A, Lowe M. Acceptance and commitment therapy as a novel treatment for eating disorders: an initial test of efficacy and mediation. Behav Modif. 2013 Jul;37(4):459-89. doi: 10.1177/0145445513478633. Epub 2013 Mar 8. PMID 23475153
- [Background] Sharp WG, Jaquess DL, Morton JF, Herzinger CV. Pediatric feeding disorders: a quantitative synthesis of treatment outcomes. Clin Child Fam Psychol Rev. 2010 Dec;13(4):348-65. doi: 10.1007/s10567-010-0079-7. PMID 20844951
- [Background] Couturier J, Kimber M, Szatmari P. Efficacy of family-based treatment for adolescents with eating disorders: a systematic review and meta-analysis. Int J Eat Disord. 2013 Jan;46(1):3-11. doi: 10.1002/eat.22042. Epub 2012 Jul 23. PMID 22821753
- [Background] Arcelus J, Mitchell AJ, Wales J, Nielsen S. Mortality rates in patients with anorexia nervosa and other eating disorders. A meta-analysis of 36 studies. Arch Gen Psychiatry. 2011 Jul;68(7):724-31. doi: 10.1001/archgenpsychiatry.2011.74. PMID 21727255
- [Background] Davies H, Fox J, Naumann U, Treasure J, Schmidt U, Tchanturia K. Cognitive remediation and emotion skills training for anorexia nervosa: an observational study using neuropsychological outcomes. Eur Eat Disord Rev. 2012 May;20(3):211-7. doi: 10.1002/erv.2170. Epub 2012 Mar 20. PMID 22431401
- [Background] Svaldi J, Griepenstroh J, Tuschen-Caffier B, Ehring T. Emotion regulation deficits in eating disorders: a marker of eating pathology or general psychopathology? Psychiatry Res. 2012 May 15;197(1-2):103-11. doi: 10.1016/j.psychres.2011.11.009. Epub 2012 Mar 7. PMID 22401969
- [Background] Lattimore P, Mead BR, Irwin L, Grice L, Carson R, Malinowski P. 'I can't accept that feeling': Relationships between interoceptive awareness, mindfulness and eating disorder symptoms in females with, and at-risk of an eating disorder. Psychiatry Res. 2017 Jan;247:163-171. doi: 10.1016/j.psychres.2016.11.022. Epub 2016 Nov 16. PMID 27915166
- [Background] Lavender JM, Wonderlich SA, Engel SG, Gordon KH, Kaye WH, Mitchell JE. Dimensions of emotion dysregulation in anorexia nervosa and bulimia nervosa: A conceptual review of the empirical literature. Clin Psychol Rev. 2015 Aug;40:111-22. doi: 10.1016/j.cpr.2015.05.010. Epub 2015 Jun 6. PMID 26112760
- [Background] Linardon J, Fairburn CG, Fitzsimmons-Craft EE, Wilfley DE, Brennan L. The empirical status of the third-wave behaviour therapies for the treatment of eating disorders: A systematic review. Clin Psychol Rev. 2017 Dec;58:125-140. doi: 10.1016/j.cpr.2017.10.005. Epub 2017 Oct 23. PMID 29089145
- [Background] Haeyen S, van Hooren S, van der Veld W, Hutschemaekers G. Efficacy of Art Therapy in Individuals With Personality Disorders Cluster B/C: A Randomized Controlled Trial. J Pers Disord. 2018 Aug;32(4):527-542. doi: 10.1521/pedi_2017_31_312. Epub 2017 Sep 19. PMID 28926306
- [Background] Haeyen S, van Hooren S, van der Veld WM, Hutschemaekers G. Measuring the contribution of art therapy in multidisciplinary treatment of personality disorders: The construction of the Self-expression and Emotion Regulation in Art Therapy Scale (SERATS). Personal Ment Health. 2018 Feb;12(1):3-14. doi: 10.1002/pmh.1379. Epub 2017 Jul 21. PMID 28730717
- [Background] van den Broek, E., Keulen-de Vos, M., & Bernstein, D. P. (2011). Arts therapies and schema focused therapy: A pilot study. The Arts in Psychotherapy, 38(5), 325-332.
- [Background] Lock J, Fitzpatrick KK, Agras WS, Weinbach N, Jo B. Feasibility Study Combining Art Therapy or Cognitive Remediation Therapy with Family-based Treatment for Adolescent Anorexia Nervosa. Eur Eat Disord Rev. 2018 Jan;26(1):62-68. doi: 10.1002/erv.2571. Epub 2017 Nov 20. PMID 29152825
- [Background] Holmqvist G, Lundqvist Persson C. Is there evidence for the use of art therapy in treatment of psychosomatic disorders, eating disorders and crisis? A comparative study of two different systems for evaluation. Scand J Psychol. 2012 Feb;53(1):47-53. doi: 10.1111/j.1467-9450.2011.00923.x. Epub 2011 Oct 25. PMID 22023072
- [Background] Gatta, M., Gallo, C., & Vianello, M. (2014). Art therapy groups for adolescents with personality disorders. The Arts in Psychotherapy, 41(1), 1-6.
- [Background] Slayton, S. C., D'Archer, J., & Kaplan, F. (2010). Outcome studies on the efficacy of art therapy: A review of findings. Art therapy, 27(3), 108-118.
- [Background] Stuckey HL, Nobel J. The connection between art, healing, and public health: a review of current literature. Am J Public Health. 2010 Feb;100(2):254-63. doi: 10.2105/AJPH.2008.156497. Epub 2009 Dec 17. PMID 20019311
- [Background] Van Lith, T. (2016). Art therapy in mental health: A systematic review of approaches and practices. The Arts in Psychotherapy, 47, 9-22.
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment, 26(1), 41-54
- [Background] Garnefski, N., & Kraaij, V. (2007). The cognitive emotion regulation questionnaire. European Journal of Psychological Assessment, 23(3), 141-149.
- [Background] Garner, D. M. (2004). Eating disorder inventory-3 (EDI-3). Professional manual. Odessa, FL: Psychological Assessment Resources.